CLINICAL TRIAL: NCT00948168
Title: 6-Months Exenatide and Glucose Homeostasis Determinants in Type 2 Diabetic Patients
Brief Title: Effect of Exenatide on Glucose Homeostasis Determinants in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Service d'Endocrinologie et Nutrition, Cliniques universitaires St-Luc, Brussels
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-DIAB-01
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM; exenatide; HbA1c; weight; waist circumference; insulin sensitivity; beta-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: exenatide (Byetta) — all patients receive 5 then 10 µg exenatide subcutaneously BID for 6 months

SUMMARY:
The purpose of this study is to determine in type 2 diabetic patients in secondary failure to combined oral therapy whether, besides improvement in glycemic control, addition of exenatide, a new drug introduced to treat diabetes before addition of insulin to current therapy, over 6 months is associated with improvement in beta-cell function, insulin sensitivity following 24-hours discontinuation of the drug.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes subjects
* 40 to 80 years
* body mass index (BMI) between 25 and 40 kg/m²
* baseline glycated haemoglobin (HbA1c) > 7.0 %, despite a maximally-tolerated combined oral therapy with a BCF stimulant (sulfonylurea or repaglinide) plus metformin

Exclusion Criteria:

* previous or current use of glitazone
* previous use of systemic glucocorticoids, weight-reducing drug(s) such as sibutramine
* previous exposure to GLP-1 receptor agonist or DPP-4 inhibitors

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Improvement in HbA1c | 6 months

SECONDARY OUTCOMES:
Non-invasive modeling of glucose homeostasis determinants, including insulin sensitivity | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires St-Luc, Brussels, Brabant, Belgium